CLINICAL TRIAL: NCT02475733
Title: A Single Blind, Randomised, Multi-centre, Active Controlled, Trial To Evaluate Safety, Tolerability, Pharmacokinetics And Efficacy Of Ceftazidime And Avibactam When Given In Combination With Metronidazole, Compared With Meropenem, In Children From 3 Months To Less Than 18 Years Of Age With Complicated Intra-abdominal Infections (cIAIs)
Brief Title: Evaluation of Safety,Pharmacokinetics and Efficacy of CAZ-AVI With Metronidazole in Children Aged 3 Months to 18 Years Old With Complicated Intra-abdominal Infections (cIAIs).
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D4280C00015; C3591004 (Other: Alias Study Number); 2014-003242-28 (EudraCT Number)
Record Dates: First submitted 2015-05-25; First posted 2015-06-19 (Estimated); Results first posted 2018-08-09 (Actual); Last update posted 2018-08-09 (Actual); Status verified 2018-07

CONDITIONS: Complicated Intra-abdominal Infections
MeSH Terms: interventions — avibactam, ceftazidime drug combination; Meropenem; Metronidazole

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CAZ-AVI and metronidazole (Experimental): CAZ-AVI to be administered every 8 hours as a 2 hour infusion (CAZ-AVI dose and frequency of IV administration will depend upon body weight and renal function) followed by metronidazole (no later than 30 minutes after CAZ-AVI infusion ) to be administered every 8 hours as 20 to 30 minutes infusion
  Interventions: Drug: Ceftazidime -avibactam; Drug: Metronidazole
- Meropenem (Active Comparator): administered every 8 hours infused over 15 to 30 minutes or up to 1 hour or infusion duration as per local guidelines.
  Interventions: Drug: Meropenem

INTERVENTIONS:
Drug: Ceftazidime -avibactam — Randomisation (3:1) to ceftazidime -avibactam plus metronidazole or meropenem treatment
  Arms: CAZ-AVI and metronidazole
Drug: Meropenem — Randomisation (3:1) to CAZ AVI plus metronidazole or meropenem treatment
  Arms: Meropenem
Drug: Metronidazole — Randomisation (3:1) to ceftazidime -avibactam plus metronidazole or meropenem treatment
  Arms: CAZ-AVI and metronidazole

SUMMARY:
This study will assess the safety , efficacy and pharmacokinetics of ceftazidime avibactam and metronidazole versus meropenem in paediatric population (from 3 months to less than 18 years of age )with complicated intra-abdominal infections (cIAIs)

DETAILED DESCRIPTION:
This is a multicentre, multinational, single blind, randomised and active controlled trial of intravenous ceftazidime avibactam in combination with metronidazole versus meropenem. Patients will receive intravenous (IV) treatment for a minimum of 72 hours (3 full days, ie, 9 doses) before having the option to switch to an oral therapy. The decision to switch to oral therapy is entirely at the Investigator's discretion, if the patient has good or sufficient clinical response, and the patient is tolerating oral fluids or food.Patients will be assessed for safety and efficacy throughout the study, and blood samples will be taken for pharmacokinetic (PK) assessment. The duration of each patient's participation in the study will be a minimum of 27 days to a maximum of 50 days after start of study treatment (defined as the time point at which first dose of study treatment is administered) at which time there will be a late follow up (LFU) assessment visit. The LFU is to be performed 20 to 35 days after the last dose of any treatment.The assessments at the test of cure (TOC) visit should be performed in person 8 to 15 days after last dose of any study drug (IV or oral). The maximum duration of IV study drug or oral switch therapy is up to Day 15.

ELIGIBILITY:
Inclusion Criteria:

1. Must be ≥3 calendar months to <18 years of age. Patients aged ≥3 calendar months to <1 year must have been born at term (defined as gestational age ≥37 weeks).
2. Written informed consent from parent(s) or other legally acceptable representative(s), and informed assent from patient (if age appropriate according to local regulations)
3. If female and has reached menarche, or has reached Tanner stage 3 development (even if not having reached menarche) (refer to Appendix E for further details on Tanner staging), the patient is authorised to participate in this clinical study if the following criteria are met:

At screening:

(i) Patient reports sexual abstinence for the prior 3 months or reports use of at least 1 of the acceptable methods of contraception, including an intrauterine device (with copper banded coil), levonorgestrel intrauterine system (eg, Mirena®), or regular medroxyprogesterone injections (Depo-Provera®); or (b) Patient agrees to initiate sexual abstinence from the time of screening until 7 days after end of treatment with study drug; and (ii) Patient is advised to avoid conception from the time of screening until 7 days after receipt of study drug and agrees not to attempt pregnancy from the time of screening until 7 days after end of treatment with study drug; and (iii) Patient is provided guidelines regarding continuation of abstinence, initiation of abstinence, or about allowed contraception; and (iv) Patient has a negative serum β-human chorionic gonadotropin (β-hCG) test just prior to study entry. Since serum tests may miss an early pregnancy, relevant menstrual history and sexual history, including methods of contraception, should be considered. Note: if the result of the serum β-hCG test cannot be obtained prior to dosing of investigational product, a patient may be enrolled on the basis of a negative urine pregnancy test, though a serum β-hCG test result must still be obtained.

4. Must, based on the judgment of the Investigator, require hospitalisation initially and antibacterial therapy for 7 to 15 days in addition to surgical intervention for the treatment of the current cIAI 5. Require surgical intervention (eg, laparotomy, laparoscopic surgery or percutaneous drainage) to manage the cIAI 6. Must have clinical evidence of cIAI as follows: (i) Pre-operative enrolment inclusion:

1. Requires surgical intervention that is expected to be completed within 24 hours of enrolment Laparotomy, laparoscopy, or percutaneous drainage
2. Evidence of a systemic inflammatory response (at least 1): Fever (defined as oral temperature >38.5°C, or equivalent to method used) or hypothermia (with a core body or rectal temperature <35°C, or equivalent to method used) Elevated white blood cells (WBC) (>15000 cells/mm3) C-reactive protein (CRP) levels (>10 mg/L)
3. Physical Findings consistent with intra-abdominal infection, such as:

   Abdominal pain and/or tenderness Localised or diffuse abdominal wall rigidity Abdominal mass
4. Intention to send specimens from the surgical intervention for culture
5. (Optional) Supportive radiologic findings of intra-abdominal infection, such as perforated intraperitoneal abscess detected on: Computed tomography (CT) scan or Magnetic resonance imaging (MRI) or Ultrasound (ii) Intra-operative/postoperative enrolment inclusion(in cases of postoperative enrolment, must be within 24 hours after the time of incision)::

Visual confirmation of intra-abdominal infection associated with peritonitis at laparotomy, laparoscopy or percutaneous drainage (to be confirmed pending feasibility); must have 1 of these diagnoses:

1. Appendiceal perforation or peri-appendiceal abscess
2. Cholecystitis with gangrenous rupture or perforation or progression of the infection beyond the gallbladder wall
3. Acute gastric or duodenal perforations, only if operated on >24 hours after singular perforation occurs
4. Traumatic perforation of the intestines, only if operated on >12 hours after perforation occurs
5. Secondary peritonitis (but not spontaneous bacterial peritonitis associated with cirrhosis and chronic ascites)

Exclusion Criteria:

1. Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study site)
2. Previous enrolment or randomisation in the present study
3. Participation in another clinical study with an investigational product (IP) during the last 30 days before the first dose of IV study drug or have previously participated in the current study or in another study of CAZ-AVI (in which an active agent was received)
4. History of hypersensitivity reactions to carbapenems, cephalosporins, penicillin, other β lactam antibiotics metronidazole or to nitroimidazole derivatives
5. Concurrent infection, that may interfere with the evaluation of response to the study antibiotics at the time of randomisation
6. Patient needs effective concomitant systemic antibacterials (oral, IV, or intramuscular) in addition to those designated in the 2 study groups (CAZ-AVI plus metronidazole group or meropenem group) (see Section 7.8)
7. Receipt of non-study systemic antibacterial drug therapy for cIAI for a continuous duration of more than 24 hours during the 72 hours preceding the first dose of IV drug, except in proven resistant organisms and/or worsening of the clinical condition for more than 24 hours. More than 2 consecutive doses are not permitted if the individual doses are expected to give >12 hours' cover (ie, giving a total cover of >24 hours.) For patients enrolled after a surgical procedure, only 1 dose of non study antibiotics is permitted postoperatively
8. Patient is considered unlikely to survive the 6 to 8 week study period
9. Patient is unlikely to respond to 7 to 15 days of treatment with antibiotics
10. Patient is receiving haemodialysis or peritoneal dialysis
11. Diagnosis of abdominal wall abscess confined to musculature of the abdominal wall or ischaemic bowel disease without perforation, traumatic bowel perforation requiring surgery within 12 hours of perforation, or perforation of gastroduodenal ulcers requiring surgery within 24 hours of perforation (these are considered situations of peritoneal soiling before the infection has become established)
12. Simple (uncomplicated), non-perforated appendicitis or gangrenous appendicitis without rupture into the peritoneal cavity identified during a surgical procedure OR presence of primary peritonitis (ie, spontaneous bacterial peritonitis) or peritonitis associated with cirrhosis or chronic ascites
13. At the time of randomisation, patient is known to have a cIAI caused by pathogens resistant to the study antimicrobials planned to be used in the study
14. Presence of any of the following clinically significant laboratory abnormalities:

    1. Haematocrit <25% or haemoglobin <8 g/dL (<80g/L , <4.9 mmol/L)
    2. Serum alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >3×the age-specific upper limit of normal (ULN), or total bilirubin >2×ULN (except known Gilbert's disease) For a) to b): unless if these values are acute and directly related to the infectious process being treated.
15. Creatinine clearance<30 mL/min /1.73 m2 calculated using the child's measured height (length) and serum creatinine within the updated "bedside" Schwartz formula (Schwartz et al, 2009):

    CrCl (mL/min/1.73m2)=0.413×height (length) (cm)/serum creatinine (mg/dL)
16. History of seizures, excluding well-documented febrile seizure of childhood
17. Any situation or condition that would make the patient, in the opinion of the Investigator, unsuitable for the study (eg, would place a patient at risk or compromise the quality of the data) or may interfere with optimal participation in the study
18. If female, currently pregnant or breast feeding

Ages: 3 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 83 (Actual)
Dates: Start 2015-08-01 (Actual); Primary Completion 2017-06-01 (Actual); Study Completion 2017-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (35):
- United States (4):
  - CHOC Children's, Orange, California
  - Rady Children's Hospital San Diego, San Diego, California
  - ProMedica Toledo Children's Hospital, Toledo, Ohio
  - The Children's Hospital at Saint Francis, Tulsa, Oklahoma
- Czechia (10):
  - Oblastni Nemocnice Kolin, a.s., Nemocnice Stredoceskeho Kraje, Detske oddeleni, Kolin III
  - Lekarna Oblastni Nemocnice Kolin, a.s., Kolin III
  - Krajska zdravotni, a.s. - Nemocnice Most, o.z., Detske a dorostove oddeleni, Most
  - Lekarna Nemocnice Most, o.z., Most
  - Fakultni Nemocnice Ostrava - Klinika Detskeho Lekarstvi, Ostrava - Poruba
  - Lekarna Fakultni Nemocnice Ostrava, Ostrava - Poruba
  - Lekarna Thomayerovy Nemocnice, Praha 4 - Krc
  - Thomayerova Nemocnice, Klinika detske chirurgie a traumatologie 3.LF UK a TN, Praha 4 - Krc
  - Lekarna Nemocnice Strakonice, Strakonice
  - Nemocnice Strakonice, a.s. - Detske oddeleni, Strakonice
- Greece (2):
  - General Children's Hospital of Athens "P. & A.Kyriakou", Athens, Attica
  - General Hospital of Thessaloniki "Hippokratio", Thessaloniki, Macedonia
- Hungary (5):
  - Semmelweis Egyetem, II. sz. Gyermekgyogyaszati Klinika, Budapest
  - Kanizsai Dorottya Korhaz, Csecsemo es Gyermekgyogyaszati Osztaly, Nagykanizsa
  - Pecsi Tudomanyegyetem, AOK, Klinikai Kozpont, Gyermekgyogyaszati Klinika, Pécs
  - Szegedi Tudomanyegyetem, Szent-Gyorgyi Albert Klinikai Kozpont, Szeged
  - Tolna Megyei Balassa Janos Korhaz, Gyermekgyogyaszati Osztaly, Szekszárd
- Uniwersytecki Szpital Dzieciecy w Lublinie, Lublin, Poland
- Spitalul Clinic de Urgenta pentru Copii "Sf. Maria" Iasi, Sectia Chirurgie Pediatrica II, Iași, Romania
- State Budgetary Educational Institution of Higher Professional Education, Smolensk, Smolensk Oblast, Russia
- Spain (5):
  - Hospital Universitario Germans Trias i Pujol, Badalona, Barcelona
  - Hospital de Sant Joan de Deu, Esplugues de Llobregat, Barcelona
  - Hospital Clinico San Carlos, Madrid
  - Hospital Universitario Fundacion Jimenez Diaz, Madrid
  - Hospital Universitario y Politecnico la Fe, Valencia
- Taiwan (3):
  - Kaohsiung Veterans General Hospital, Kaohsiung City
  - Taichung Veterans General Hospital, Taichung
  - Department of Pediatrics, Mackay Memorial Hospital, Taipei
- Turkey (Türkiye) (3):
  - Cukurova Universitesi Tip Fakultesi Balcali Hastanesi, Adana
  - Eskisehir Osmangazi Universitesi Saglik Uygulama ve Arastirma Hastanesi, Eskişehir
  - Celal Bayar Universitesi Hafsa Sultan Hastanesi, Manisa

REFERENCES:
- [Derived] Franzese RC, McFadyen L, Watson KJ, Riccobene T, Carrothers TJ, Vourvahis M, Chan PLS, Raber S, Bradley JS, Lovern M. Population Pharmacokinetic Modeling and Probability of Pharmacodynamic Target Attainment for Ceftazidime-Avibactam in Pediatric Patients Aged 3 Months and Older. Clin Pharmacol Ther. 2022 Mar;111(3):635-645. doi: 10.1002/cpt.2460. Epub 2021 Nov 22. PMID 34687548
- [Derived] Bradley JS, Broadhurst H, Cheng K, Mendez M, Newell P, Prchlik M, Stone GG, Talley AK, Tawadrous M, Wajsbrot D, Yates K, Zuzova A, Gardner A. Safety and Efficacy of Ceftazidime-Avibactam Plus Metronidazole in the Treatment of Children >/=3 Months to <18 Years With Complicated Intra-Abdominal Infection: Results From a Phase 2, Randomized, Controlled Trial. Pediatr Infect Dis J. 2019 Aug;38(8):816-824. doi: 10.1097/INF.0000000000002392. PMID 31306396

RESULTS

PARTICIPANT FLOW:
Groups:
- Ceftazidime- Avibactam (CAZ-AVI) Plus Metronidazole: Participants with Creatinine clearance(CrCL) >=50 milliliter per minute (mL/min) received 10 milligram per kilogram (mg/kg) intravenous(IV) infusion of metronidazole over 20 to 30 minutes along with 2 hour IV infusion of CAZ/AVI in following manner: 1)Age 6 to less than(<)18 years: 2000 mg CAZ/500 mg AVI (body weight >=40 kg), 50 mg/kg CAZ/12.5 mg/kg AVI (body weight <40 kg), 2) Age 6 months to <6 years: 50 mg/kg CAZ/12.5 mg/kg AVI, 3)Age 3 months to <6 months: 40 mg/kg CAZ/10 mg/kg AVI. Both infusions were administered to participants every 8 hours for a minimum of 72 hours and up to a maximum duration of 15 days. Dose of CAZ-AVI was drops below to 50% if CrCl of participant drops below to 50mL/min, and participant was removed from study therapy, if CrCl decreased below 30mL/min. After having 72 hours of IV treatment, participants had option to switch to an oral therapy at investigator's discretion.
- Meropenem: Participants received 15 to 30 minutes IV infusion of meropenem 20 mg/kg every 8 hours for a minimum of 72 hours and up to a maximum duration of 15 days. After having 72 hours of IV treatment, participants had option to switch to an oral therapy at the investigator's discretion.
Period: Overall Study
Arm/Group | Ceftazidime- Avibactam (CAZ-AVI) Plus Metronidazole | Meropenem
Started | 61 | 22
Completed | 59 | 22
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) analysis set included all participants who had been assigned a randomized treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Ceftazidime- Avibactam (CAZ-AVI) Plus Metronidazole | Meropenem | Total
Number analyzed (Participants) | 61 | 22 | 83
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.4 (3.64) | 9.7 (3.97) | 10.2 (3.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 13 | 30
  Male | 44 | 9 | 53
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 1 | 13
  Not Hispanic or Latino | 49 | 21 | 70
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 7 | 4 | 11
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 53 | 16 | 69
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged in-patient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent AEs were events between first dose of study drug and up to late follow-up (LFU) visit (20 to 35 days after last dose of study treatment [IV or oral]) that were absent before treatment or that worsened relative to pretreatment state. AEs included both SAE and non-SAE.
Time Frame: Baseline until the LFU visit (up to a maximum study duration of 50 days)
Population: Safety analysis set included all randomized participants who received any amount of IV study medication (CAZ-AVI plus Metronidazole or Meropenem).
Measure: Number; unit: percentage of participants
Arm/Group | Ceftazidime- Avibactam (CAZ-AVI) Plus Metronidazole | Meropenem
Number analyzed (Participants) | 61 | 22
percentage of participants
  AEs | 52.5 | 59.1
  SAEs | 8.2 | 4.5

2. Primary Outcome: Percentage of Participants With Cephalosporin Class Effects and Additional Adverse Events (AEs)
Description: Percentage of participants with Cephalosporin class effects (defined as adverse event of special interest (AEoSI) within the safety topics (ST) of hypersensitivity/anaphylaxis) and additional AEs (which included AEs of seizures, diarrhea, renal disorder, and liver disorder relevant to the cephalosporin class within the ST and AEs with preferred term in the system organ class of nervous system disorder system organ class based on MedDRA 20.0) were reported in this outcome measure.
Time Frame: Baseline until the LFU visit (up to a maximum study duration of 50 days)
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Ceftazidime- Avibactam (CAZ-AVI) Plus Metronidazole | Meropenem
Number analyzed (Participants) | 61 | 22
percentage of participants
  AE in the ST of Diarrhea | 1.6 | 0
  AEoSI in the ST of Hypersensitivity/Anaphylaxis | 4.9 | 13.6
  AE in the ST of Liver Disorder | 0 | 0
  AE in the ST of Renal Disorder | 0 | 0
  AEs with PTs in the Nervous System Disorder SOC | 1.6 | 4.5
  AE of seizure | 0 | 0

3. Primary Outcome: Change From Baseline in Pulse Rate at End of Intravenous Therapy (EOIV) Visit
Description: EOIV visit occurred within 24 hours after completion of last infusion of the study drug.
Time Frame: Baseline, EOIV visit (anytime from Day 4 up to 16)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Ceftazidime- Avibactam (CAZ-AVI) Plus Metronidazole | Meropenem
Number analyzed (Participants) | 61 | 22
beats per minute
  Baseline | 102.1 (17.07) | 103.0 (23.31)
  Change at EOIV: number analyzed (Participants) | 60 | 22
  Change at EOIV | -15.2 (20.45) | -15.4 (21.74)

4. Primary Outcome: Change From Baseline in Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP) at End of Intravenous Therapy (EOIV) Visit
Description: EOIV visit occurred within 24 hours after completion of last infusion of the study drug.
Time Frame: Baseline, EOIV visit (anytime from Day 4 up to 16)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: millimeter of mercury (mmHg)
Arm/Group | Ceftazidime- Avibactam (CAZ-AVI) Plus Metronidazole | Meropenem
Number analyzed (Participants) | 61 | 22
millimeter of mercury (mmHg)
  SBP: Baseline: number analyzed (Participants) | 60 | 22
  SBP: Baseline | 109.7 (13.90) | 111.6 (13.06)
  SBP: Change at EOIV: number analyzed (Participants) | 59 | 22
  SBP: Change at EOIV | -4.0 (12.32) | -6.0 (13.66)
  DBP: Baseline: number analyzed (Participants) | 60 | 22
  DBP: Baseline | 63.5 (10.36) | 63.1 (13.51)
  DBP: Change at EOIV: number analyzed (Participants) | 59 | 22
  DBP: Change at EOIV | 1.3 (11.99) | -2.8 (14.14)

5. Primary Outcome: Change From Baseline in Respiratory Rate at End of Intravenous Therapy (EOIV) Visit
Description: EOIV visit occurred within 24 hours after completion of last infusion of the study drug.
Time Frame: Baseline, EOIV visit (anytime from Day 4 up to 16)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: breaths per minute
Arm/Group | Ceftazidime- Avibactam (CAZ-AVI) Plus Metronidazole | Meropenem
Number analyzed (Participants) | 61 | 22
breaths per minute
  Baseline: number analyzed (Participants) | 58 | 21
  Baseline | 22.4 (5.02) | 22.9 (5.79)
  Change at EOIV: number analyzed (Participants) | 56 | 21
  Change at EOIV | -1.3 (4.57) | -1.3 (4.44)

6. Primary Outcome: Change From Baseline in Body Weight at End of Intravenous Therapy (EOIV) Visit
Description: EOIV visit occurred within 24 hours after completion of last infusion of the study drug.
Time Frame: Baseline, EOIV visit (anytime from Day 4 up to 16)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Ceftazidime- Avibactam (CAZ-AVI) Plus Metronidazole | Meropenem
Number analyzed (Participants) | 61 | 22
kilograms
  Baseline | 40.58 (16.286) | 38.35 (16.685)
  Change at EOIV: number analyzed (Participants) | 56 | 20
  Change at EOIV | -0.38 (1.442) | -1.06 (1.490)

7. Primary Outcome: Change From Baseline in Body Temperature at End of Intravenous Therapy (EOIV) Visit
Description: EOIV visit occurred within 24 hours after completion of last infusion of the study drug.
Time Frame: Baseline, EOIV visit (anytime from Day 4 up to 16)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: degree Celsius
Arm/Group | Ceftazidime- Avibactam (CAZ-AVI) Plus Metronidazole | Meropenem
Number analyzed (Participants) | 61 | 22
degree Celsius
  Baseline: number analyzed (Participants) | 60 | 22
  Baseline | 37.35 (1.035) | 37.16 (0.914)
  Change at EOIV: number analyzed (Participants) | 59 | 22
  Change at EOIV | -0.78 (0.987) | -0.60 (0.780)

8. Primary Outcome: Percentage of Participants With Abnormal Physical Examination Findings at End of Intravenous Therapy (EOIV) Visit
Description: Physical examination included an assessment of the following: general appearance, skin, head and neck (including ears, eyes, nose and throat), lymph nodes, thyroid, respiratory system, cardiovascular system, abdomen, musculoskeletal system (including spine and extremities), and neurological system. Participants with new or aggravated abnormal physical examination findings with regard to baseline findings were reported. Abnormality in physical examinations were based on blinded observer's discretion. EOIV visit occurred within 24 hours after completion of last infusion of the study drug.
Time Frame: EOIV visit (anytime from Day 4 up to 16)
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Ceftazidime- Avibactam (CAZ-AVI) Plus Metronidazole | Meropenem
Number analyzed (Participants) | 61 | 22
percentage of participants
  Abdomen | 6.6 | 18.2
  Cardiovascular System | 0 | 0
  General Appearance | 1.6 | 0
  Head and Neck | 0 | 0
  Lymph Nodes | 0 | 0
  Musculoskeletal System | 0 | 0
  Neurological System | 0 | 0
  Respiratory System | 3.3 | 0
  Skin | 1.6 | 0
  Thyroid | 0 | 0

9. Primary Outcome: Percentage of Participants With Potentially Clinically Significant Abnormalities in Laboratory Parameters
Description: Criteria for potentially clinically significant laboratory abnormalities: Chemistry (calcium: <0.7*lower limit of normal range [LLN] and >30 percent decrease from baseline [DFB]; alanine aminotransferase [ALT]: >3*upper limit of normal range [ULN] and >300 percent IFB; alanine aminotransferase [AST]: >3*ULN and >300 percent IFB) and hematology (platelets: >2*ULN and >100 percent IFB). LFU visit occurred within 20 to 35 days after last dose of study treatment (IV or oral).
Time Frame: Baseline until the LFU visit (up to a maximum study duration of 50 days)
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Ceftazidime- Avibactam (CAZ-AVI) Plus Metronidazole | Meropenem
Number analyzed (Participants) | 61 | 22
percentage of participants
  Chemistry: Calcium: number analyzed (Participants) | 53 | 21
  Chemistry: Calcium | 1.9 | 0
  Chemistry: ALT: number analyzed (Participants) | 59 | 22
  Chemistry: ALT | 1.7 | 0
  Chemistry: AST: number analyzed (Participants) | 55 | 21
  Chemistry: AST | 1.8 | 0
  Hematology: Platelets: number analyzed (Participants) | 60 | 22
  Hematology: Platelets | 3.3 | 0

10. Primary Outcome: Percentage of Participants With Electrocardiogram (ECG) Parameter QTcF: > 450, >480 and >500 Millisecond (ms)
Description: ECG parameters included maximum QT intervals using Fridericia's correction (QTcF). Maximum QTcF >450 millisecond (ms); maximum QTcF >480 ms; and maximum QTcF >500 ms. EOIV visit occurred within 24 hours after completion of last infusion of the study drug.
Time Frame: Baseline until the EOIV visit (anytime from Day 4 to 16)
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Ceftazidime- Avibactam (CAZ-AVI) Plus Metronidazole | Meropenem
Number analyzed (Participants) | 61 | 22
percentage of participants
  Maximum QTcF Interval : >450 ms | 1.6 | 4.5
  Maximum QTcF Interval : >480 ms | 1.6 | 4.5
  Maximum QTcF Interval : >500 ms | 0 | 4.5

11. Primary Outcome: Percentage of Participants With Creatinine Clearance (CrCl) at Day 7
Description: CrCl is a measure of glomerular filtration rate (GMFR), an index of kidney function. It is the volume of blood plasma that is cleared of creatinine by the kidneys per unit time. Percentage of participants with CrCl in the following categories were reported: <30 mL/min/1.73 m^2, >=30 to <50 mL/min/1.73 m^2, >=50 mL/min/1.73 m^2 to <80 mL/min/1.73 m^2, and >=80 mL/min/1.73 m^2.
Time Frame: Day 7
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Ceftazidime- Avibactam (CAZ-AVI) Plus Metronidazole | Meropenem
Number analyzed (Participants) | 61 | 22
percentage of participants
  CrCl: <30mL/min/1.73 m^2 | 0 | 0
  CrCl: >=30 to <50mL/min/1.73 m^2 | 0 | 0
  CrCl: >=50 to <80mL/min/1.73 m^2 | 0 | 0
  CrCl: >=80mL/min/1.73 m^2 | 50.8 | 59.1

12. Primary Outcome: Percentage of Participants With Creatinine Clearance (CrCl) at End of Intravenous Therapy (EOIV) Visit
Description: CrCl is a measure of GMFR, an index of kidney function. It is the volume of blood plasma that is cleared of creatinine by the kidneys per unit time. Percentage of participants with CrCl in the following categories were reported: <30 mL/min/1.73 m^2, >=30 to <50 mL/min/1.73 m^2, >=50 mL/min/1.73 m^2 to <80 mL/min/1.73 m^2, and >=80 mL/min/1.73 m^2. EOIV visit occurred within 24 hours after completion of last infusion of the study drug.
Time Frame: EOIV visit (anytime from Day 4 up to 16)
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Ceftazidime- Avibactam (CAZ-AVI) Plus Metronidazole | Meropenem
Number analyzed (Participants) | 61 | 22
percentage of participants
  CrCl: <30mL/min/1.73 m^2 | 0 | 0
  CrCl: >=30 to <50mL/min/1.73 m^2 | 0 | 0
  CrCl: >=50 to <80mL/min/1.73 m^2 | 0 | 0
  CrCl: >=80mL/min/1.73 m^2 | 82.0 | 81.8

13. Primary Outcome: Percentage of Participants With Creatinine Clearance (CrCl) at Test of Cure (TOC) Visit
Description: CrCl is a measure of GMFR, an index of kidney function. It is the volume of blood plasma that is cleared of creatinine by the kidneys per unit time. Percentage of participants with CrCl in the following categories were reported: <30 mL/min/1.73 m^2, >=30 to <50 mL/min/1.73 m^2, >=50 mL/min/1.73 m^2 to <80 mL/min/1.73 m^2, and >=80 mL/min/1.73 m^2. TOC visit occurred within 8 to 15 days after last dose of any study drug (IV or oral).
Time Frame: TOC visit (up to a maximum study duration of 50 days)
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Ceftazidime- Avibactam (CAZ-AVI) Plus Metronidazole | Meropenem
Number analyzed (Participants) | 61 | 22
percentage of participants
  CrCl: <30mL/min/1.73 m^2 | 0 | 0
  CrCl: >=30 to <50mL/min/1.73 m^2 | 0 | 0
  CrCl: >=50 to <80mL/min/1.73 m^2 | 3.3 | 0
  CrCl: >=80mL/min/1.73 m^2 | 42.6 | 59.1

14. Primary Outcome: Percentage of Participants With Creatinine Clearance (CrCl) at Late Follow-up (LFU) Visit
Description: CrCl is a measure of GMFR, an index of kidney function. It is the volume of blood plasma that is cleared of creatinine by the kidneys per unit time. Percentage of participants with CrCl in the following categories were reported: <30 mL/min/1.73 m^2, >=30 to <50 mL/min/1.73 m^2, >=50 mL/min/1.73 m^2 to <80 mL/min/1.73 m^2, and >=80 mL/min/1.73 m^2. LFU visit occurred within 20 to 35 days after last dose of study treatment (IV or oral).
Time Frame: LFU visit (up to a maximum study duration of 50 days)
Population: Safety analysis set included all randomized participants who received any amount of IV study medication.
Measure: Number; unit: percentage of participants
Arm/Group | Ceftazidime- Avibactam (CAZ-AVI) Plus Metronidazole | Meropenem
Number analyzed (Participants) | 61 | 22
percentage of participants
  CrCl: <30mL/min/1.73 m^2 | 0 | 0
  CrCl: >=30 to <50mL/min/1.73 m^2 | 0 | 0
  CrCl: >=50 to <80mL/min/1.73 m^2 | 1.6 | 0
  CrCl: >=80mL/min/1.73 m^2 | 6.6 | 9.1

15. Secondary Outcome: Plasma Concentrations of Ceftazidime and Avibactam
Time Frame: 15, 30-90, 300-360 minutes post-dose on Day 3
Population: PK analysis set included all randomized participants who received any amount of study medication and had at least 1 CAZ and/ or AVI plasma measurement available. This outcome measure was not planned to be analyzed for meropenem receiving cohorts, as pre-specified in protocol.
Measure: Geometric Mean (Standard Deviation); unit: nanogram per milliliter
Arm/Group | Ceftazidime- Avibactam (CAZ-AVI) Plus Metronidazole
Number analyzed (Participants) | 60
nanogram per milliliter
  Ceftazidime: 15 minute post-dose on Day 3: number analyzed (Participants) | 59
  Ceftazidime: 15 minute post-dose on Day 3 | 63565.5 (236761.80)
  Ceftazidime: 30-90 minute post-dose on Day 3 | 38048.0 (19810.95)
  Ceftazidime:300-360minute post-dose on Day 3 | 4603.0 (10308.96)
  Avibactam: 15 minute post-dose on Day 3: number analyzed (Participants) | 59
  Avibactam: 15 minute post-dose on Day 3 | 12186.2 (55720.44)
  Avibactam: 30-90 minute post-dose on Day 3 | 6548.6 (4437.55)
  Avibactam: 300-360 minute post-dose on Day 3 | 821.5 (1968.21)

16. Secondary Outcome: Percentage of Participants With Favorable Clinical Response (CR) at End of 72 Hours Treatment: Intent-to-treat (ITT) Analysis Population
Description: Favorable CR was defined as resolution of all acute signs and symptoms of complicated intra- abdominal infection (cIAIs), or improvement to such an extent that no further antimicrobial therapy was required, or improvement but not enough to switch to oral therapy and still on IV study drug at end of 72 hours and had met following criterion: absence of new signs and symptoms, improvement in at least 1 symptom/sign (fever, pain, tenderness, elevated White Blood Cells [WBCs], elevated c-reactive protein) from baseline and no worsening symptom/sign.
Time Frame: End of 72 hours study drug treatment on Day 1
Population: ITT analysis population included all participants who had been assigned a randomized treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ceftazidime- Avibactam (CAZ-AVI) Plus Metronidazole | Meropenem
Number analyzed (Participants) | 61 | 22
percentage of participants | 93.4 [85.2 to 97.7] | 90.9 [73.9 to 98.1]

17. Secondary Outcome: Percentage of Participants With Favorable Clinical Response (CR) at End of Intravenous Therapy (EOIV) Visit: Intent-to-treat (ITT) Analysis Population
Description: Favorable CR was resolution of all acute signs and symptoms of cIAI or improvement to such an extent that no further antimicrobial therapy was required, or improvement in participants who had switch to oral therapy and met the following criterion: afebrile (temperature <=38.0°C) for at least 24 hours, absence of new and improvement in at least 1 symptom or sign (fever, pain, tenderness, elevated WBCs, elevated c-reative-protein) from baseline and worsening of none. EOIV visit occurred within 24 hours after completion of last infusion of the study drug.
Time Frame: EOIV visit (anytime from Day 4 up to 16)
Population: ITT analysis population included all participants who had been assigned a randomized treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ceftazidime- Avibactam (CAZ-AVI) Plus Metronidazole | Meropenem
Number analyzed (Participants) | 61 | 22
percentage of participants | 96.7 [89.9 to 99.3] | 100 [89.3 to 100]

18. Secondary Outcome: Percentage of Participants With Favorable Clinical Response (CR) at End of Treatment (EOT) Visit: Intent-to-treat (ITT) Analysis Population
Description: Favorable CR was resolution of all acute signs and symptoms of cIAI, or improvement to such an extent that no further antimicrobial therapy was required. EOT visit occurred within 48 hours after completion of the last dose of oral switch therapy or at time of premature discontinuation/early withdrawal from study (if on oral switch therapy).
Time Frame: EOT visit (up to Day 17)
Population: ITT analysis population included all participants who had been assigned a randomized treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ceftazidime- Avibactam (CAZ-AVI) Plus Metronidazole | Meropenem
Number analyzed (Participants) | 61 | 22
percentage of participants | 91.8 [83.0 to 96.8] | 100 [89.3 to 100]

19. Secondary Outcome: Percentage of Participants With Favorable Clinical Response (CR) at Test of Cure (TOC) Visit: Intent-to-treat (ITT) Analysis Population
Description: Favorable CR was resolution of all acute signs and symptoms of cIAI, or improvement to such an extent that no further antimicrobial therapy was required. TOC visit occurred within 8 to 15 days after last dose of any study drug (IV or oral).
Time Frame: TOC visit (up to a maximum study duration of 50 days)
Population: ITT analysis population included all participants who had been assigned a randomized treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ceftazidime- Avibactam (CAZ-AVI) Plus Metronidazole | Meropenem
Number analyzed (Participants) | 61 | 22
percentage of participants | 91.8 [83.0 to 96.8] | 95.5 [80.7 to 99.5]

20. Secondary Outcome: Percentage of Participants With Favorable Clinical Response (CR): Clinically Evaluable (CE) Analysis Population
Description: Favorable CR was resolution of all acute signs and symptoms of cIAI, or improvement to such an extent that no further antimicrobial therapy was required, or improvement in participants who had switch to oral therapy and met the following criterion: afebrile (temperature <=38.0°C) for at least 24 hours, absence of new and improvement in at least 1 symptom or sign (fever, pain, tenderness, elevated WBCs, elevated c-reative-protein) from baseline and worsening of none. EOIV visit occurred within 24 hours after completion of last infusion of the study drug. EOT visit occurred within 48 hours after completion of last dose of oral switch therapy or at time of premature discontinuation/early withdrawal from study (if on oral switch therapy). TOC visit occurred within 8 to 15 days after last dose of any study drug (IV or oral).
Time Frame: End of 72 hours study drug treatment on Day 1, EOIV (anytime from Day 4 up to 16), EOT visit (up to Day 17) and TOC visit (up to a maximum study duration of 50 days)
Population: CE analysis population included randomized participants with cIAI who received study medication for >=48h and clinical failure or clinical failure with treatment limiting AE and participants with >=72h treatment and favorable clinicial response.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ceftazidime- Avibactam (CAZ-AVI) Plus Metronidazole | Meropenem
Number analyzed (Participants) | 56 | 20
percentage of participants
  End 72 hours study medication: number analyzed (Participants) | 49 | 20
  End 72 hours study medication | 98.0 [90.9 to 99.8] | 95.0 [78.9 to 99.5]
  EOIV: number analyzed (Participants) | 54 | 20
  EOIV | 98.1 [91.7 to 99.8] | 100 [88.3 to 100]
  EOT: number analyzed (Participants) | 52 | 20
  EOT | 94.2 [85.4 to 98.3] | 100 [88.3 to 100]
  TOC | 92.9 [83.9 to 97.5] | 95.0 [78.9 to 99.5]

21. Secondary Outcome: Percentage of Participants With Favorable Microbiological Response: Microbiological Intent-to-treat (Micro-ITT) Population
Description: Favorable microbiological response was achieved when all baseline pathogens were eradicated or presumed eradicated based on investigator's discretion. EOIV visit occurred within 24 hours after completion of last infusion of the study drug. EOT visit occurred within 48 hours after completion of last dose of oral switch therapy or at time of premature discontinuation/early withdrawal from study if on oral switch therapy (which occurred within the maximum study treatment duration of 15 days). EOIV visit occurred within 24 hours after completion of last infusion of the study drug. TOC visit occurred within 8 to 15 days after last dose of any study drug (IV or oral). LFU visit occurred within 20 to 35 days after last dose of study treatment (IV or oral).
Time Frame: EOIV visit (Day 4 up to 16), EOT visit (up to Day 17), TOC visit (up to a maximum study duration of 50 days) and LFU visit (up to a maximum study duration of 50 days)
Population: Micro-ITT analysis population included all randomized participants who had a baseline pathogen known to cause cIAI.
Measure: Number; unit: percentage of participants
Arm/Group | Ceftazidime- Avibactam (CAZ-AVI) Plus Metronidazole | Meropenem
Number analyzed (Participants) | 50 | 19
percentage of participants
  EOIV | 96.0 | 100
  EOT | 90.0 | 100
  TOC | 90.0 | 94.7
  LFU | 90.0 | 94.7

22. Secondary Outcome: Percentage of Participants With Favorable Microbiological Response: Microbiologically Evaluable (ME) Population
Description: Favorable microbiological response was achieved when all baseline pathogens were eradicated or presumed eradicated based on investigator's discretion. EOIV visit occurred within 24 hours after completion of last infusion of the study drug. EOT visit occurred within 48 hours after completion of last dose of oral switch therapy or at time of premature discontinuation/early withdrawal from study if on oral switch therapy (which occurred within the maximum study treatment duration of 15 days). TOC visit occurred within 8 to 15 days after last dose of any study drug (IV or oral). LFU visit occurred within 20 to 35 days after last dose of study treatment (IV or oral).
Time Frame: as for outcome 21
Population: ME analysis population included randomized participants with cIAI who received study medication for >=48h and clinical failure or clinical failure with treatment limiting AE and participants with >=72h treatment and favorable microbiological response.
Measure: Number; unit: percentage of participants
Arm/Group | Ceftazidime- Avibactam (CAZ-AVI) Plus Metronidazole | Meropenem
Number analyzed (Participants) | 40 | 15
percentage of participants
  EOIV | 97.5 | 100
  EOT: number analyzed (Participants) | 36 | 15
  EOT | 91.7 | 100
  TOC | 90.0 | 93.3
  LFU: number analyzed (Participants) | 37 | 14
  LFU | 89.2 | 92.9

23. Secondary Outcome: Percentage of Participants With Clinical Relapse at Late Follow-up (LFU) Visit: Clinically Evaluable (CE) Population
Description: A participant was said to have clinical relapse if met either 1 of the following criteria: reappearance or worsening of signs and symptoms of cIAI that required further antimicrobial therapy and/or surgery, or death after TOC in which cIAI was contributory. LFU visit occurred within 20 to 35 days after last dose of study treatment (IV or oral).
Time Frame: LFU visit (up to a maximum study duration of 50 days)
Population: CE analysis population included randomized participants with cIAI who received study medication for >=48h and clinical failure or clinical failure with treatment limiting AE and participants with >=72h treatment and favorable clinicial response. Here, number of participants analyzed=participants who were evaluable for this measure.
Measure: Number; unit: percentage of participants
Arm/Group | Ceftazidime- Avibactam (CAZ-AVI) Plus Metronidazole | Meropenem
Number analyzed (Participants) | 48 | 18
percentage of participants | 0 | 0

24. Secondary Outcome: Percentage of Participants With Clinical Relapse at Late Follow-up (LFU) Visit: Microbiologically Evaluable (ME) Population
Description: A participant was said to have clinical relapse if me either 1 of the following criteria: reappearance or worsening of signs and symptoms of cIAI that required further antimicrobial therapy and/or surgery, or death after TOC in which cIAI was contributory. LFU visit occurred within 20 to 35 days after last dose of study treatment (IV or oral).
Time Frame: LFU visit (up to a maximum study duration of 50 days)
Population: ME analysis population included randomized participants with cIAI who received study medication for >=48 h and clinical failure or clinical failure with treatment limiting AE and participants with >=72 h treatment and favorable microbiological response. Here, number of participants analyzed=participants who were evaluable for this measure.
Measure: Number; unit: percentage of participants
Arm/Group | Ceftazidime- Avibactam (CAZ-AVI) Plus Metronidazole | Meropenem
Number analyzed (Participants) | 37 | 14
percentage of participants | 0 | 0

25. Secondary Outcome: Percentage of Participants With Emergent Infections: Microbiological Intent-to-treat (Micro-ITT) Population
Description: Emergent infections were categorized as super infections and new infections. Superinfection: An intra-abdominal culture identified pathogen other than a baseline pathogen during the course of active treatment with study therapy along with worsening signs and symptoms of infection requiring alternative antimicrobial therapy. New infection: An intra-abdominal culture identified pathogen other than a baseline pathogen at any time after study treatment had finished along with worsening signs and symptoms of infection requiring alternative antimicrobial therapy. Participants with any (super infections or new infections) of the infections were reported.
Time Frame: Baseline up to 50 days
Population: Micro-ITT analysis population included all randomized participants who had a baseline pathogen known to cause cIAI.
Measure: Number; unit: percentage of participants
Arm/Group | Ceftazidime- Avibactam (CAZ-AVI) Plus Metronidazole | Meropenem
Number analyzed (Participants) | 50 | 19
percentage of participants | 0 | 0

26. Secondary Outcome: Percentage of Participants With Emergent Infections at Test of Cure (TOC) Visit: Microbiologically Evaluable Population
Description: Emergent Infections was an intra-abdominal culture identified pathogen other than a baseline pathogen during the course of active treatment with study therapy along with worsening signs and symptoms of infection requiring alternative antimicrobial therapy, new infection was an intra-abdominal culture identified pathogen other than a baseline pathogen at any time after study treatment has finished along with worsening signs and symptoms of infection requiring alternative antimicrobial therapy. TOC visit occurred within 8 to 15 days after last dose of any study drug (IV or oral). Participants with any (super infections or new infections) of the infections were reported.
Time Frame: TOC visit (up to a maximum study duration of 50 days)
Population: ME analysis population included randomized participants with cIAI who received study medication for >=48 h and clinical failure or clinical failure with treatment limiting AE and participants with >=72 h treatment and favorable microbiological response.
Measure: Number; unit: percentage of participants
Arm/Group | Ceftazidime- Avibactam (CAZ-AVI) Plus Metronidazole | Meropenem
Number analyzed (Participants) | 40 | 15
percentage of participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline until the LFU visit (up to a maximum study duration of 50 days)
Description: Same event may appear as both an AE and SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another, or a participant may have experienced both a serious and non-serious event.
Arm/Group | Ceftazidime- Avibactam (CAZ-AVI) Plus Metronidazole | Meropenem
All-Cause Mortality (participants affected / at risk) | 0/61 | 0/22
Serious Adverse Events (participants affected / at risk) | 5/61 | 1/22
Other Adverse Events (participants affected / at risk) | 14/61 | 6/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ceftazidime- Avibactam (CAZ-AVI) Plus Metronidazole (N=61) | Meropenem (N=22)
Ileus (Gastrointestinal disorders) | 1 | 1
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Large intestine perforation (Gastrointestinal disorders) | 1 | 0
Postoperative ileus (Injury, poisoning and procedural complications) | 1 | 0
Renal colic (Renal and urinary disorders) | 1 | 0
Urethral meatus stenosis (Renal and urinary disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ceftazidime- Avibactam (CAZ-AVI) Plus Metronidazole (N=61) | Meropenem (N=22)
Abdominal pain (Gastrointestinal disorders) | 0 | 2
Vomiting (Gastrointestinal disorders) | 9 | 2
Infusion site phlebitis (General disorders) | 4 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2017-03-07): https://cdn.clinicaltrials.gov/large-docs/33/NCT02475733/Prot_000.pdf
  • Statistical Analysis Plan (2017-08-24): https://cdn.clinicaltrials.gov/large-docs/33/NCT02475733/SAP_001.pdf